CLINICAL TRIAL: NCT03513029
Title: Clinical Investigation of the VytronUS Ablation System for Treatment of Symptomatic Drug-refractory Paroxysmal Atrial Fibrillation
Acronym: VITAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VytronUS, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 980-08694-00
Record Dates: First submitted 2018-04-27; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: PAF; atrial fibrillation; ablation; low intensity collimated ultrasound
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Device (Experimental): VytronUS Ablation System
  Interventions: Device: VytronUS Ablation System

INTERVENTIONS:
Device: VytronUS Ablation System — Catheter Ablation for Paroxysmal Atrial Fibrillation

SUMMARY:
VITAL is a prospective, single arm, multicenter, interventional study to evaluate the safety and effectiveness of the VytronUS Ablation System (VAS) for the treatment of symptomatic paroxysmal atrial fibrillation (PAF) using low intensity collimated ultrasound (LICU) for imaging and ablation.

DETAILED DESCRIPTION:
Patients undergoing elective catheter ablation for symptomatic PAF who are refractory or intolerant to at least one antiarrhythmic drug (Class I-IV) will be screened for enrollment. Patients who meet the study entry criteria and sign the patient informed consent form will be enrolled and treated consistent with the 2012 Heart Rhythm Society (HRS)/European Heart Rhythm Association (EHRA)/European Cardiac Arrhythmia Society (ECAS) Expert Consensus Statement on Catheter and Surgical Ablation for Atrial Fibrillation. Eligible patients will receive treatment with the VAS including ultrasound imaging of the left atrium and cardiac ablation to electrically isolate the pulmonary veins.

Up to 100 patients will be enrolled at up to 10 sites in Europe (EU) and in the United States (US).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* History of symptomatic recurrent paroxysmal atrial fibrillation (PAF) in the prior year, defined by:

  1. Two or more symptomatic AF episodes lasting greater than 30 seconds duration that self-terminate and lasting no more than 7 continuous days. An episode of AF ≤ 48 hours duration terminated with electrical or pharmacologic cardioversion counts as a paroxysmal atrial fibrillation episode.
  2. At least one episode of paroxysmal atrial fibrillation (PAF) documented on 12-lead ECG, event monitor, or telemetry monitor in the prior year
* Paroxysmal atrial fibrillation refractory to at least one Beta Blocker, Calcium Channel Blocker, or Class I or Class III anti-arrhythmic drug (AAD).
* Subject is indicated for a pulmonary vein ablation according to society guidelines or investigational site practice.
* Subject is able and willing to give informed consent.
* Willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full duration of the study

Exclusion Criteria:

* Prior LA ablation or surgery
* Persistent, longstanding persistent, or permanent AF
* AF secondary to electrolyte imbalance, thyroid disease or reversible or non-cardiac cause
* NYHA Class III or IV congestive heart failure
* Rheumatic heart disease
* Atrial myxoma
* LVEF <40% measured by acceptable cardiac testing (e.g. TTE, TEE)
* Anteroposterior LA diameter >5.5cm or <3.5cm by TTE, CT or MRI
* Presence of intracardiac thrombus (including a known history of thrombus) within 30 days prior to the index ablation procedure
* Presence of pulmonary vein stent(s)
* Presence of pre-existing pulmonary narrowing or pulmonary vein stenosis greater than 70%
* Presence of pre-existing pericardial effusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety: Incidence of early-onset serious adverse events | 7 days or discharge, whichever is sooner
  Incidence of early-onset serious adverse events
Primary Effectiveness: Acute success and chronic freedom from AF, AFL or AT | 12 months
  Acute success and chronic freedom from AF, AFL or AT

SECONDARY OUTCOMES:
Secondary Safety: All serious adverse events | 12 months
  All serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No